CLINICAL TRIAL: NCT04848766
Title: Comparison of De-escalation Treatment Strategy After Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrome
Brief Title: IPD Meta-analysis of De-escalation Treatment Strategy After PCI in ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: St. Antonius Hospital (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: De-escal-meta
Record Dates: First submitted 2021-04-10; First posted 2021-04-19 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: percutaneous coronary intervention; dual antiplatelet therapy; de-escalation
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- De-escalation treatment group: Patients diagnosed as acute coronary syndrome, and who receive de-escalation antiplatelet therapy after percutaneous coronary intervention
  Interventions: Drug: De-escalation Treatment Strategy of dual antiplatelet therapy
- Conventional treatment group: Patients diagnosed as acute coronary syndrome, and who receive conventional (non-de-escalation) antiplatelet therapy after percutaneous coronary intervention

INTERVENTIONS:
Drug: De-escalation Treatment Strategy of dual antiplatelet therapy — Patients receive de-escalation treatment of dual antiplatelet therapy after percutaneous coronary intervention
  Groups: De-escalation treatment group

SUMMARY:
We will perform a systemic review of previously published data and an updated patient-level meta-analysis of studies, including the most recent publications. PubMed, EMBASE, Cochrane Central Register of Controlled Trials, the United States National Institutes of Health registry of clinical trials, and relevant websites were searched for pertinent published studies.

DETAILED DESCRIPTION:
This is an individual patient-level data meta-analysis (IPD Meta-analysis). This study population was incorporated from studies that were previoiusly published.

We will perform a systemic review of previously published data and an updated patient-level meta-analysis of studies, including the most recent publications. PubMed, EMBASE, Cochrane Central Register of Controlled Trials, the United States National Institutes of Health registry of clinical trials, and relevant websites were searched for pertinent published studies. The electronic search strategy was complemented by manual examination of references cited by included articles, recent reviews, editorials, and meta-analyses. No restrictions were imposed on language, study period, or sample size. The search keywords include "acute coronary syndrome", "ACS", "primary", "percutaneous coronary intervention", "PCI", "de-escalation", "guided", "guide", "antiplatelet", "P2Y12 inhibitor", "P2Y12", "dual antiplatelet therapy", "DAPT".

Articles were included when they met the following prespecified criteria: (1) included the ACS patients who underwent PCI with drug-eluting stent (DES); (2) maintained DAPT for 1 year; (3) de-escalation strategy of DAPT was clearly defined; (4) clinical outcomes, including ischemic and bleeding events, were clearly reported; (5) randomized controlled trials were considered for inclusion. Two independent investigators screened titles and abstracts, identified duplicated studies, performed full-article reviews, and determined the study inclusion. The third investigator supervised the searching process and adjudicated all the disagreements.

After selecting eligible RCTs, we will incorporate all known randomized controlled trials requesting individual patient data from the principal investigator of each trial.

ELIGIBILITY:
This study is a meta-analysis of previously published studies. Therefore, the eligibility criteria may be diverse according to the individual studies.

--------------------------

Inclusion Criteria:

* Subject must have clinical diagnosis of acute coronary syndrome

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Prasugrel, Ticagrelor

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical and cerebral events (NACCE) | 1 year after intervention
  composite of all-cause death, myocardial infarction, coronary revascularization, stroke and major bleeding.

SECONDARY OUTCOMES:
Composite endpoint of Major adverse cardiovascular outcomes | 1 year after intervention
  all-cause mortality, myocardial infarction, coronary revascularization, stroke
Major Bleeding outcome defined by the Bleeding Academic Research Consortium (BARC) criteria | 1 year after intervention
  Bleeding outcomes, defined by the Bleeding Academic Research Consortium criteria
Individual components of the primary outcome | 1 year after intervention
  all-cause mortality
Individual components of the primary outcome | 1 year after intervention
  cardiovascular mortality
Individual components of the primary outcome | 1 year after intervention
  non-cardiovascular mortality
Individual components of the primary outcome | 1 year after intervention
  myocardial infarction
Individual components of the primary outcome | 1 year after intervention
  stroke
Individual components of the primary outcome | 1 year after intervention
  any coronary revascularization
Individual components of the primary outcome | 1 year after intervention
  any bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Woo Park, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be decided after discussed with the principle investigators of each study.